CLINICAL TRIAL: NCT04306068
Title: Efficacy of an Intervention by Plyometrics in the Ankle Stabilizers in the Improvement of the Balance in Salsa Dancers From 18 to 25 Years. A Randomized Clinical Study.
Brief Title: Plyometrics in the Ankle Stabilizing Muscles in Improving Balance in Ballerinas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 coronavirus pandemic
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DANCE
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Balance; Distorted
Keywords: Balance; Plyometrics; Dance; Stability; Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Athletes included in the experimental group will perform a plyometric exercise protocol. Each session will consist of a 4-station circuit with 1 minute rest between each station and 30 seconds between sets
  Interventions: Other: Plyometric protocol
- Control group (No Intervention): Athletes included in the control group will follow their usual warm-up routine.

INTERVENTIONS:
Other: Plyometric protocol — Each session will last 20 minutes, with 2 sessions a week, over a period of 5 weeks. The intervention will last 20 minutes, which consists of a 4-station circuit.
  Exercise 1: jump on the rope, with your feet together at a moderate pace. Exercise 2: In standing with hands on the hip and hip flexion (one foot in front). Knee flexion and dorsal ankle flexion, with straight trunk. Alternate legs.
  Exercise 3: box jump (jump on the box with both feet at the same time). Exercise 4: depth jumps from box to antoher box (jump on the box with both feet at the same time and when falling, immediately jump to the other box).
  1 minute with 30 seconds between sets.
  Arms: Experimental group

SUMMARY:
Balance is essential for successful dance performance. The effort of salsa dancers is given by the levels of stability, produced by the muscular activation of lower limbs.

The objective of the study is to assess the effectiveness of an intervention of plyometric exercises in the improvement of balance in salsa dancers from 18 to 25 years.

Randomized clinical study. 40 dancers will be randomized to the two study groups: experimental (application of plyometric exercise protocol) and control (without intervention). The treatment will last 5 weeks, with 2 weekly sessions of 25 minutes each. The dependent variables will be: equilibrium (measured with star excursion balance). The sample distribution will be calculated using the Kolmogorov-Smirnof test. The changes after each evaluation will be calculated with the t-student test. With an ANOVA of repeated measures, the intra and intersubject effect will be observed. The effect size will be obtained with Cohen's formula.

It is expected to see improvement in the stability of the ankle and the level of balance in the dancers.

ELIGIBILITY:
Inclusion Criteria:

* Dancers
* Female
* From 18 to 25 years
* With more than a year of dance practice
* And without musculoskeletal injury at the time of starting the study.

Exclusion Criteria:

* Subjects who do not attend all training sessions
* Pregnant women or intending to remain in state during the study period
* Have not signed the informed consent

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The Star excursion balance test will be used. Before performing the test, the movements will be explained. The test will be calculated in 3 directions with three tapes 140cm long and with a goniometer the subsequent sections of 135º from the previous section will be calculated, and 45º between the subsequent sections.
  Participants will start standing with both feet with the midpoint on the intersection mark in the center of the grid. They will be instructed to keep their hands on their hips, their heads facing forward at all times and keeping their feet flat on the floor trying to reach as far as possible in all three directions. The range will be measured by marking the tape with a pen and then measured with a measurement quote.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain